CLINICAL TRIAL: NCT06828107
Title: A Prospective, Non-randomized, Sequentially-enrolled, Multi-center, Phase II Study to Evaluate the SENSE Device's Ability to Detect Traumatic Brain Injury
Brief Title: A Study to Evaluate the SENSE Device's Ability to Detect TBI
Acronym: SENSE-007
Status: Recruiting | Type: Observational
Sponsor: Sense Diagnostics, LLC (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SENSE-007; TP230368 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
Keywords: SENSE Device
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- TBI patients with intracranial bleeding: 50 patients with TBI with intracranial bleeding
  Interventions: Device: SENSE device
- TBI patients without intracranial bleeding: 50 patients with TBI without intracranial bleeding
  Interventions: Device: SENSE device
- Control subjects with normal brain health: 50 control subjects with normal brain health
  Interventions: Device: SENSE device

INTERVENTIONS:
Device: SENSE device — The SENSE Device transmits a low power tailored electro-magnetic (EM) pulse in the radio-frequency range across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage and/or cerebral edema.

SUMMARY:
The study population will consist of 3 mutually-exclusive sets of patients and subjects:

* TBI patients with intracranial bleeding
* TBI patients without intracranial bleeding
* Control subjects with normal brain health.

Research subjects ages 22 and older will be enrolled. All TBI patients must be monitored with the SENSE Device within 6 hours of a diagnostic head CT scan ordered by a treating clinician and within 24 hours of injury.

DETAILED DESCRIPTION:
This study is a phase II, prospective, non-randomized, multi-center, within patient and between-group comparison of the SENSE Device and the standard diagnostic test, head CT scan, in patients with a diagnosis of TBI with or without intracranial bleeding (defined as epidural hemorrhage, subdural hemorrhage, subarachnoid hemorrhage, and/or traumatic contusions/intraparenchymal hemorrhage) and subjects with normal brain health for the detection of intracranial hemorrhages.

The following pair-wise comparisons will be performed to address the following research questions:

Is there a difference in the agreement between the head CT scan and the SENSE Device for detecting intracranial bleeding in patients with TBI? Patients with TBI with intracranial bleeding vs. Patients with TBI without intracranial bleeding (Objective no. 1)

Is there a difference in the false positive rate for the presence of bleeding between patients with TBI without intracranial bleeding and control subjects with normal brain health? Patients with TBI without intracranial bleeding vs. control subjects (Objective no. 1)

This study is a phase II, prospective, non-randomized, multi-center, within patient and between-group comparison of the SENSE Device and the standard diagnostic test, head CT scan, in patients with a diagnosis of TBI with or without intracranial bleeding (defined as epidural hemorrhage, subdural hemorrhage, subarachnoid hemorrhage, and/or traumatic contusions/intraparenchymal hemorrhage) and subjects with normal brain health for the detection of intracranial hemorrhages.

The following pair-wise comparisons will be performed to address the following research questions:

Is there a difference in the agreement between the head CT scan and the SENSE Device for detecting intracranial bleeding in patients with TBI? Patients with TBI with intracranial bleeding vs. Patients with TBI without intracranial bleeding (Objective no. 1)

Is there a difference in the false positive rate for the presence of bleeding between patients with TBI without intracranial bleeding and control subjects with normal brain health? Patients with TBI without intracranial bleeding vs. control subjects (Objective no. 1)

A separate set of evaluations will be performed, pooling the patients with TBI without intracranial bleeding on initial head CT and the control subjects. The agreements between the SENSE Device and the head CT scan will be compared between these 2 groups:

Patients with TBI with intracranial bleeding vs. Subjects without intracranial bleeding (both TBI patients and control subjects).

All subjects who meet eligibility criteria should be enrolled. One-hundred (100) patients with TBI (50 with intracranial hemorrhage and 50 without intracranial hemorrhage) will be enrolled to determine whether the SENSE Device can distinguish patients with TBI with intracranial hemorrhage from those without intracranial hemorrhage. Fifty (50) control subjects with normal brain health will be enrolled for comparison to patients with TBI. All subjects will be monitored for 15 minutes with the SENSE Device. Control subjects will not undergo any brain imaging. Control subjects will be enrolled based on symptom evaluation at the time of enrollment.

A core radiology lab using independent readers will verify the presence or absence of intracranial hemorrhage and cerebral edema for all scans and will quantify hemorrhage and edema volumes using computer-assisted analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female adults age 22 and older

  * Patients with TBI who have a head CT scan obtained in the mobile stroke unit, emergency department, or hospital, ordered by a treating clinician OR control subjects with normal brain health.
  * For patients with traumatic intracranial hemorrhage, blood is visible on ≥ 3 consecutive axial CT slices.
  * Signed written informed consent by study subject or, if subject is unable, by subject's next of kin or legally authorized representative.
  * Willingness and ability to comply with schedule for study procedures.

Exclusion Criteria:

* • Female patients who are pregnant or lactating.

  * SENSE Device is unable to be placed within 6 hours of a standard of care head CT and within 24 hours of injury.
  * Open skull fracture (closed skull fracture is not an exclusion).
  * Metallic intracranial clip, coil, or device (such as metallic ICP monitor).
  * Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for the SENSE Device monitoring or study participation or may confound the outcome of the study.
  * Planned placement of an intraventricular catheter prior to study enrollment.
  * Planned intracranial surgery prior to study enrollment.
  * Current participation in a medical or surgical interventional clinical trial.
  * Use of continuous EEG monitoring at the time of enrollment.
  * Clinical uncertainty about the presence or absence of hemorrhage on the enrolling head CT.
  * Control subjects with normal brain health will have no known history of seizure, stroke, brain tumor, TBI requiring emergency room evaluation, concussion within the previous 6 months, hydrocephalus, intracranial vascular malformation, other structural brain disease, or intracranial surgery. Benign headache disorders (e.g. migraine headache, tension headache), and mild concussion > 6 months prior to enrollment are not exclusions.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 3 mutually-exclusive sets of patients and subjects:
  * TBI patients with intracranial bleeding
  * TBI patients without intracranial bleeding
  * Control subjects with normal brain health.
  Research subjects ages 22 and older will be enrolled. All TBI patients must be monitored with the SENSE Device within 6 hours of a diagnostic head CT scan ordered by a treating clinician and within 24 hours of injury.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 12 months
  The SENSE output for each patient will be classified as showing intracranial hemorrhage or no intracranial hemorrhage for each study CT with corresponding SENSE data. The SENSE output will be compared with the gold standard (CT scan result) to determine the accuracy of the SENSE Device as classifying TBI patients with and without intracranial hemorrhage correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Jason McMullan, MD, Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - University of Florida, Gainesville, Florida
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - UT Houston, Houston, Texas
  - UTSA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
We have not made a determination yet as a company